CLINICAL TRIAL: NCT01571557
Title: A Safety and Efficacy Study to Assess OZURDEX® in Patients With Macular Oedema Secondary to Retinal Vein Occlusion (RVO)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/RET/011
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OZURDEX®: OZURDEX® (dexamethasone 700 ug intravitreal implant) administered according to standard of care.
  Interventions: Drug: dexamethasone 700 ug intravitreal implant

INTERVENTIONS:
Drug: dexamethasone 700 ug intravitreal implant — dexamethasone 700 ug intravitreal implant administered according to standard of care.
  Other Names: OZURDEX®

SUMMARY:
This study will evaluate the relationship between time since onset of macular oedema symptoms and the achievement of vision gain in patients prescribed OZURDEX®. All care and diagnostic procedures provided are at the discretion of the participating physicians according to their clinical judgment and local standard of medical care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of macular edema following retinal vein occlusion
* Prescribed OZURDEX®

Exclusion Criteria:

* Previous treatment with OZURDEX®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with macular oedema due to retinal vein occlusion
Sampling Method: Non-Probability Sample
Enrollment: 573 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Berlin, Germany

REFERENCES:
- [Background] Augustin AJ, Holz FG, Haritoglou C, Mayer WJ, Bopp S, Scheuerle AF, Maier M, Sekundo W, Sandner D, Shirlaw A, Hattenbach LO. Retrospective, observational study in patients receiving a dexamethasone intravitreal implant 0.7 mg for macular oedema secondary to retinal vein occlusion. Ophthalmologica. 2015;233(1):18-26. doi: 10.1159/000368840. Epub 2014 Dec 5. PMID 25503473

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OZURDEX®
Started | 573
Completed | 573
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OZURDEX®
Number analyzed (Participants) | 573
Age, Customized [Count of Participants; unit: Participants]
  31 to 40 years | 4
  41 to 50 years | 13
  51 to 60 years | 69
  61 to 70 years | 127
  71 to 80 years | 235
  81 to 90 years | 119
  91 to 100 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286
  Male | 287

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured in the study eye following each injection of OZURDEX® using the Snellen eye chart. BCVA measurements expressed in Snellen fractions are converted to logMAR units and the approximate Early Treatment Diabetic Retinopathy Study (ETDRS) letter score is based on the formula: approximate ETDRS letters=85+50 x log10 (Snellen fraction). The converted scores are "approximate ETDRS letters" to distinguish the scores from visual acuity measurements obtained using the ETDRS chart. One line on the EDTRS equals 5 ETDRS points. The lower the number of letters read correctly on the eye chart (lower number on the decimal scale) the worse the vision (or visual acuity). The higher the number of letters read correctly (higher number on the decimal scale), the better the vision (or visual acuity). A positive number change from baseline in the number of letters read means vision has improved and a negative number change from baseline means vision has worsened.
Time Frame: Baseline, Week 12
Population: All enrolled patients with complete data at this time point
Measure: Mean (Standard Deviation); unit: Approximate EDTRS Letters
Arm/Group | OZURDEX®
Number analyzed (Participants) | 351
Approximate EDTRS Letters
  Baseline | 52.431 (18.929)
  Change from Baseline at Week 12 | 7.774 (14.986)

2. Secondary Outcome: Percentage of Patients With an Increase of ≥2 Lines From Baseline BCVA in the Study Eye
Description: BCVA is measured in the study eye following each injection of OZURDEX® using the Snellen eye chart. BCVA measurements expressed in Snellen fractions are converted to logMAR units and the approximate ETDRS letter score is based on the formula: approximate ETDRS letters=85+50 x log10 (Snellen fraction). The converted scores are "approximate ETDRS letters" to distinguish the scores from visual acuity measurements obtained using the ETDRS chart. One line on the EDTRS equals 5 ETDRS points. The lower the number of letters read correctly on the eye chart (lower number on the decimal scale) the worse the vision (or visual acuity). An increase of 2 letters or more indicates an improvement in BCVA.
Time Frame: Baseline, 48 Weeks
Population: All enrolled patients
Measure: Number; unit: Percentage of Patients
Arm/Group | OZURDEX®
Number analyzed (Participants) | 573
Percentage of Patients | 46.60

3. Secondary Outcome: Percentage of Patients With an Increase of ≥3 Lines From Baseline BCVA in the Study Eye
Description: BCVA is measured in the study eye following each injection of OZURDEX® using the Snellen eye chart. BCVA measurements expressed in Snellen fractions are converted to logMAR units and the approximate ETDRS letter score is based on the formula: approximate ETDRS letters=85+50 x log10 (Snellen fraction). The converted scores are "approximate ETDRS letters" to distinguish the scores from visual acuity measurements obtained using the ETDRS chart. One line on the EDTRS equals 5 ETDRS points. The lower the number of letters read correctly on the eye chart (lower number on the decimal scale) the worse the vision (or visual acuity). An increase of 3 letters or more indicates an improvement in BCVA.
Time Frame: Baseline, 48 Weeks
Population: All enrolled patients
Measure: Number; unit: Percentage of Patients
Arm/Group | OZURDEX®
Number analyzed (Participants) | 573
Percentage of Patients | 36.47

4. Secondary Outcome: Mean Change From Baseline in Central Retinal Thickness
Description: Retinal thickness is assessed by optical coherence tomography (OCT) in the study eye. The retina is the light-sensitive part of the eye. OCT is a laser-based, noninvasive, diagnostic system providing high-resolution, three-dimensional images of the retina. A negative mean change from baseline indicates an improvement and a positive mean change from baseline indicates a worsening.
Time Frame: Baseline, Week 24
Population: All enrolled patients with complete data at this time point
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | OZURDEX®
Number analyzed (Participants) | 343
micrometers (μm)
  Baseline | 501.18 (169.30)
  Change from Baseline at Week 24 (N=138) | -61.75 (192.28)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from the time of the first OZURDEX® injection through the final follow-up visit for each patient.
Description: All enrolled patients were used to assess AEs and SAEs.
Arm/Group | OZURDEX®
Serious Adverse Events (participants affected / at risk) | 1/573
Other Adverse Events (participants affected / at risk) | 33/573
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OZURDEX® (N=573)
Glaucoma (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OZURDEX® (N=573)
Intraocular Pressure Increased (Eye disorders) | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.